CLINICAL TRIAL: NCT02668250
Title: The OPTI-AGED Study : Influence of a Multi-parametric Optimization Strategy for General Anesthesia on Postoperative Morbidity and Mortality in Elderly Patients. A Randomized, Multicentre, Prospective Controlled Study
Brief Title: Influence of a Multi-parametric Optimization Strategy for General Anesthesia on Postoperative Morbidity and Mortality
Acronym: OPTI-AGED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1508190; ANSM (Other: 2016-A00667-44)
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Coronary; Ischemic; Arrhythmias, Cardiac; Heart Failure; Peripheral Vascular Diseases; Dementia; Stroke; Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Alcoholism; Cancer; Diabetes; Renal Insufficiency
MeSH Terms: conditions — Ischemia; Arrhythmias, Cardiac; Heart Failure; Peripheral Vascular Diseases; Dementia; Stroke; Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Alcoholism; Neoplasms; Diabetes Mellitus; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : OPTI-AGED (Experimental): The OPTI-AGED group will receive a combined optimization strategy of anesthesia concerning hemodynamic, ventilation, and depth of anesthesia.
  Interventions: Procedure: OPTI-AGED
- Control Group : (Active Comparator): The control group will not benefit from the OPTI-AGED intervention but patients will receive the usual care.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: OPTI-AGED — OPTI-AGED is composed of a multi-parametric optimization strategy.
  Arms: Experimental group : OPTI-AGED
Procedure: Usual Care — Patients receive the usual care.
  Arms: Control Group :

SUMMARY:
With the increasing aging population demographics and life expectancies, the number of very elderly patients undergoing surgery is rising. Elderly patients constitute an increasingly large proportion of the high-risk surgical group.

Cardiac complications and postoperative pulmonary complications are equally prevalent and contribute similarly to morbidity, mortality, and length of hospital stay. Specific optimization strategy of general anesthesia has been tested in high-risk patients undergoing major surgery to improve outcomes.

Our hypothesis is that a combined optimization strategy of anesthesia concerning hemodynamic, ventilation, and depth of anesthesia may improve short- and long- term outcome in elderly undergoing high risk surgery.

DETAILED DESCRIPTION:
The population is expanding and aging. With the increasing aging population demographics and life expectancies, the number of very elderly patients (age ≥ 75) undergoing surgery is rising. Elderly patients constitute an increasingly large proportion of the high-risk surgical group. In 2010, patients aged 75 yrs and over represented only 2.1% of patients undergoing high risk surgery in France (PMSI database), but concentrated 27% of in-hospital deaths.

Cardiac complications and postoperative pulmonary complications are equally prevalent and contribute similarly to morbidity, mortality, and length of hospital stay. Specific optimization strategy of general anesthesia has been tested in high-risk patients undergoing major surgery to improve outcomes. Meta-analyses have demonstrated that goal directed hemodynamic therapy significantly reduced mortality and surgical complications in high-risk patients. A lung-protective ventilation strategy in high-risk patients undergoing major abdominal surgery was associated with improved clinical outcome. Retrospective studies indicated that a combination of excessive depth of anesthesia, hypotension and low anesthesia requirement resulted in increased mortality. These approaches of peroperative care remain discussed in the literature and have also to be incorporated in the common clinical practice. Moreover, few of these reviews performed a sensitive analysis in the elderly.

Whether a multi-parametric optimization strategy of anesthesia including several specific interventions will impact the short-term postoperative major morbidity and mortality in elderly is not known. The addition of depth of anesthesia monitoring to hemodynamic monitoring and goal directed hemodynamic therapy may improve tissue perfusion by reducing hemodynamic side effects of anesthetic agents, particularly in elderly where the therapeutic window of these agents is reduced. The effects of low protective ventilation may also by additive to the previous measures by reducing the perioperative build-up of oxygen debt. Our hypothesis is that a combined optimization strategy of anesthesia concerning hemodynamic, ventilation, and depth of anesthesia may improve short- and long- term outcome in elderly undergoing high risk surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 75 years and over,
* presenting at least one of the following comorbidities: ischemic coronary disease; cardiac arrhythmia; congestive heart failure; peripheral vascular disease; dementia; stroke; chronic obstructive pulmonary disease; chronic respiratory failure; chronic alcohol abuse; active cancer; diabetes; chronic renal failure A comorbidity index will be measured by using the modified Charlson Comorbidity Index
* undergoing elective and emergency surgeries including : femoral head fracture, major intraperitoneal abdominal surgery lasting > 90 min (excluding elective cholecystectomy, abdominal wall surgery), vascular surgery (excluding venous surgery and fistula creation)
* Patient's or patient's relative signed consent form
* Affiliation to French social assurance system

Exclusion Criteria:

* Acute heart failure and acute coronary syndrome
* Acute respiratory failure, pneumonia
* Septic shock
* Delirium
* Acute stroke
* Evolutive neuromuscular disorder
* Thoracic surgery, combined abdominal and thoracic surgery
* Surgery performed under exclusive regional anesthesia
* Patients under tutorship or curatorship
* Refusal to participate

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2495 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Incidence of a composite of mortality or major postoperative morbidity. | Day 30
  One or more of major postoperative complications : acute kidney injury (defined by Kidney disease : improving Global Outcomes (KDIGO) stage 1 or higher), acute myocardial infarction, heart failure, stroke, development of sepsisand septic shock, acute respiratory failure requiring non-invasive ventilation or intubation, delirium) will be reported in the source folder of the patients, and the mortality will be also focused. The goal of this study is to decrease this incidence.

CONTACTS AND LOCATIONS:
Overall Officials: MOLLIEX Serge, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (29):
- France (29):
  - CHU Amiens - Picardie, Amiens
  - CHU CAEN, Caen
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Médipôle Lyon - Villeurbanne, Décines-Charpieu
  - Chu Dijon, Dijon
  - Chu Grenoble, Grenoble
  - CHRU Lille - Salengro, Lille
  - CHU LILLE - Huriez, Lille
  - CHU LYON, Lyon
  - Lyon Sud - CHU, Lyon
  - Chu Marseille La Timone, Marseille
  - Chu Marseille Nord, Marseille
  - Chu Montpellier, Montpellier
  - Chu Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU NICE, Nice
  - Chu Nimes, Nîmes
  - Ch Paris Beaujon, Paris
  - Ch Paris Bichat, Paris
  - Ch Paris Pitie Salpetriere, Paris
  - Ch Paris Saint Antoine, Paris
  - Ch Saint Louis-Lariboisiere, Paris
  - Chu Poitiers, Poitiers
  - Chu Rennes, Rennes
  - Chu Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Hopital Central Strasbourg, Strasbourg
  - Hopital Hautepierre Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molliex S, Passot S, Futier E, Bonnefoi M, Rancon F, Lemanach Y, Pereira B. Stepped wedge cluster randomised controlled trial to assess the effectiveness of an optimisation strategy for general anaesthesia on postoperative morbidity and mortality in elderly patients (the OPTI-AGED study): a study protocol. BMJ Open. 2018 Jun 19;8(6):e021053. doi: 10.1136/bmjopen-2017-021053. PMID 29921685